CLINICAL TRIAL: NCT05332574
Title: A Phase I/II, First-in-Human, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of a Trispecific EGFR/cMET/cMET Antibody GB263T in Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC) and Other Solid Tumors
Brief Title: A Safety, Tolerability, PK and Preliminary Activity Study of GB263T in Advanced NSCLC and Other Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB263T-FIH001
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-03

CONDITIONS: NSCLC; Other Solid Tumors
Keywords: NSCLC; Phase 1/2; GB263T; EGFR/cMET/cMET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB263T (Experimental): Experimental: GB263T
  Interventions: Biological: GB263T

INTERVENTIONS:
Biological: GB263T — Participants will receive IV infusions of GB263T at increased dose level until maximum tolerated dose is reached or all planned doses are administered. Participants will receive GB263T at predefined dose levels and frequency, based upon observed safety and protocol defined criteria. The duration of each treatment cycle is 28 days.

SUMMARY:
This is a Phase 1/2 study of GB263T in participants with advanced NSCLC and other solid tumor. The study will consist of a dose-escalation and expansion stage to determine RP2D (Phase 1), and an extension stage (Phase 2) where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Subjects with histologically or cytologically confirmed metastatic or unresectable advanced NSCLC or other solid tumors who have progressed on prior standard therapy, have been intolerant to prior standard therapy, or have refused all other currently available therapeutic options.
3. Subjects must have evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. ECOG PS 0-1.
5. An expected survival time is ≥3 months.
6. Adequate organ function.
7. Subjects in Phase II must agree to provide pre-treatment tumor tissue samples.

Exclusion Criteria:

1. Subjects who have had prior chemotherapy, targeted cancer therapy, immunotherapy, or any investigational anti-cancer treatment within 2 weeks or five half-lives of the treatment (whichever is longer), prior to the first administration of the study drug.
2. Toxicity (excluding alopecia, peripheral neuropathy, and hypothyroidism) that did not return to class 0 or class 1 of NCI CTCAE V5.0 from prior antitumor therapy prior to the first administration of the study drug.
3. Prior radical radiation therapy completed within 4 weeks prior to the first administration of the study drug.
4. Subjects with untreated symptomatic brain metastases.
5. History of interstitial lung disease (ILD).
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
7. Received live virus vaccination within 30 days of first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs | Screening up to follow-up (30 [+7] days after the last dose)
DLT in Phase I | During Cycle 1 (up to 28 days)
ORR in Phase II | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose)

SECONDARY OUTCOMES:
Cmax | At predefined intervals up to 449 days
Tmax | At predefined intervals up to 449 days
AUC0-last | At predefined intervals up to 449 days
AUC0-τ | At predefined intervals up to 449 days
t1/2 | At predefined intervals up to 449 days
Cmin | At predefined intervals up to 449 days
Rac_Cmax | At predefined intervals up to 449 days
Rac_AUC0-τ | At predefined intervals up to 449 days
ADA | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose)
PFS | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose
DOR | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose)
CBR | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose)
OS | Up to End of Treatment (EOT) Follow Up Period (30 [+7] days after the last dose)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Genesis Care, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Cabrini Hospital Malvern, Malvern, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No